CLINICAL TRIAL: NCT00144066
Title: A Randomized Phase III Trial of Chemotherapy Alone Versus Chemotherapy Followed by Gefitinib in Stage IIIB/IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West Japan Thoracic Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJTOG0203
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2005-09-02 (Estimated); Status verified 2005-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Platinum Compounds; Gefitinib

INTERVENTIONS:
Drug: platinum-based chemotherapy alone (up to six cycles)
Drug: platinum-based chemotherapy followed by maintenance therapy with gefitinib

SUMMARY:
A randomized phase III trial of platinum-based chemotherapy alone versus platinum-based chemotherapy followed by maintenance therapy with gefitinib in patients with stage IIIB/IV NSCLC.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed NSCLC Stage IIIB/IV No prior treatment Measurable disease ECOG PS 0-1 Adequate organ function Age 20-74 Written informed consent

Exclusion Criteria:

Pregnancy or breast feeding Past history of drug hypersensitivity SVC syndrome Pleural or pericardial effusion that required drainage Active infection Interstitial pneumonia or active lung fibrosis Symptomatic brain metastasis Active concomitant malignancy Uncontrolled diabetes Uncontrolled heart disease

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2003-01

PRIMARY OUTCOMES:
Over all survival

SECONDARY OUTCOMES:
Time to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Toyoaki Hida, MD, PhD, Principal Investigator — West Japan Thoracic Onoclogy Group

REFERENCES:
- See also: Related Info — http://www.wjtog.org/